CLINICAL TRIAL: NCT06041360
Title: Prevalence of Peripheral Neuropathy Among Patients With Auditory Neuropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hend Abdelnasser Sayed, Resident-Audiovestibular medicine unit of ENT department-sohag hospital university, Sohag University
Other Study IDs: Soh-Med-23-07-08MS
Record Dates: First submitted 2023-09-06; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Auditory Neuropathy Spectrum Disorder,, Peripheral Neuropathy
MeSH Terms: conditions — Auditory neuropathy; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group Study group(Group1): Thirty participants of the group will meet the following criteria Inclusion criteria:
  1. Age ranges from 12 to 50 years old.
  2. Disproportionate speech recognition score (SRS) with the hearing threshold level.
  3. The auditory brainstem response (ABR) test with no waveform or, disturbed waves or, detectable wave V at high intense stimulus.
  4. The otoacoustic emission (OAE) and/or cochlear microphonic (CM) potential may be present.
  Exclusion criteria:
  While the participants who have these criteria will be excluded from the study:
  1. Consistent SRS and ABR response with hearing threshold level.
  2. Abnormal finding in brain imaging.
  3. Patients with history of diabetes and/or other causes of peripheral neuropathy.
  Interventions: Diagnostic Test: Pure tone audiometry PTA ,Speech audiometry ,Otoacoustic emission,Auditory evoked potentials including (ABR).
- Control group (Group 2): Thirty participants have the following criteria:
  1. Age and sex matched with the study group.
  2. Patients with sensorineural hearing loss with degree of hearing matched with study group
  Interventions: Diagnostic Test: Pure tone audiometry PTA ,Speech audiometry ,Otoacoustic emission,Auditory evoked potentials including (ABR).

INTERVENTIONS:
Diagnostic Test: Pure tone audiometry PTA ,Speech audiometry ,Otoacoustic emission,Auditory evoked potentials including (ABR). — Neurological tests for diagnosis of peripheral neuropathy
  Other Names: sural nerve conduction velocity (SNCV),sural nerve action potential (amplitude) (SNAP),vibration perception threshold (VPT),Michigan Neuropathy Screening

SUMMARY:
Auditory neuropathy/ dys-synchrony/ peri-synaptic audiopathy (AN) are terms used to describe a specific hearing disorder with a disturbed auditory neural response in presence of normal cochlear function. Initially reported as early as the 1970s by ( Hinchcliffe et al) after observation of the patients with normal hearing thresholds, who had difficulty to detect the sounds especially in presence of background noise . Auditory Neuropathy is characterized by five integral features that distinguish it from other types of hearing loss. These are: Variable audiometric results anywhere from normal hearing to Sensorineural hearing loss of any degree up to profound hearing loss showing unusual audiometric pattern , Preserved outer hair cells (OHCs) responses such as otoacoustic emissions (OAEs) and/or cochlear microphonics (CM) , Altered neural processing such abnormal auditory brainstem responses (ABRs) with a reduced or absent wave V , Poor speech perception with poor speech recognition score that seems out of proportion compared to their pure-tone detection thresholds. , absent stapedial reflexes to the ipsilateral and contralateral tone at a 110-dB hearing level .

In 2008 it was found that AN does not represent a single disease entity but it is a heterogeneous disease category with a wide range of hearing loss types ,etiologies , age and clinical manifestations hence the adoption of the term auditory neuropathy spectrum disorder (ANSD) by an International Newborn Hearing Screening Conference held in Italy following a comprehensive study of newborn hearing test results.

The prevalence of ANSD is variable in published studies from (0.23 to 15%) among hearing impaired individuals . Regarding the underlying etiological factors, auditory neuropathy can be congenital or acquired . AN without the involvement of the neurological system has been termed as primary auditory neuropathy (PAN).

Peripheral neuropathy is not a constant finding in all patients with this hearing disorder , AN may occur in the afferent pathway of acoustic nerve, probably accompanied by the pathological changes of efferent nerve in the olivocochlear system inside the brainstem Our study is conducted to detect the prevalence of peripheral neuropathy among patients with auditory neuropathy spectrum disorder .

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 12 to 50 years old.
* Disproportionate speech recognition score (SRS) with the hearing threshold level.
* The auditory brainstem response (ABR) test with no waveform or, disturbed waves or, detectable wave V at high intense stimulus.
* The otoacoustic emission (OAE) and/or cochlear microphonic (CM) potential may be present.

Exclusion Criteria:

* While the participants who have these criteria will be excluded from the study:

  * Consistent SRS and ABR response with hearing threshold level.
  * Abnormal finding in brain imaging.
  * Patients with history of diabetes and/or other causes of peripheral neuropathy

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Age ranges from 12 to 50 years old. Disproportionate speech recognition score (SRS) with the hearing threshold level. The auditory brainstem response (ABR) test with no waveform or, disturbed waves or, detectable wave V at high intense stimulus. The otoacoustic emission (OAE) and/or cochlear microphonic (CM) potential may be present
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Measuring the prevalence of peripheral neuropathy among patients with auditory neuropathy spectrum disorder using The Michigan neuropathy screening instrument Questionnaire and Examination | 1 year
  This measurement aims to determine the degree of disability on theses patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] De Siati RD, Rosenzweig F, Gersdorff G, Gregoire A, Rombaux P, Deggouj N. Auditory Neuropathy Spectrum Disorders: From Diagnosis to Treatment: Literature Review and Case Reports. J Clin Med. 2020 Apr 10;9(4):1074. doi: 10.3390/jcm9041074. PMID 32290039
- [Background] Gohari N, Emami SF, Mirbagheri SS, Valizadeh A, Abdollahi N, Borzuei M. The Prevalence and Causes of Auditory Neuropathy/Dys-synchrony (AN/AD) in Children with Hearing Impairment. Indian J Otolaryngol Head Neck Surg. 2019 Mar;71(1):71-75. doi: 10.1007/s12070-018-1494-1. Epub 2018 Sep 17. PMID 30906717
- [Background] Lepcha A, Chandran RK, Alexander M, Agustine AM, Thenmozhi K, Balraj A. Neurological associations in auditory neuropathy spectrum disorder: Results from a tertiary hospital in South India. Ann Indian Acad Neurol. 2015 Apr-Jun;18(2):171-80. doi: 10.4103/0972-2327.150578. PMID 26019414
- [Background] Li JK, Li W, Gao FJ, Qu SF, Hu FY, Zhang SH, Li LL, Wang ZW, Qiu Y, Wang LS, Huang J, Wu JH, Chen F. Mutation Screening of mtDNA Combined Targeted Exon Sequencing in a Cohort With Suspected Hereditary Optic Neuropathy. Transl Vis Sci Technol. 2020 Jul 8;9(8):11. doi: 10.1167/tvst.9.8.11. eCollection 2020 Jul. PMID 32855858